CLINICAL TRIAL: NCT06021119
Title: Feasibility of DPP-4 Inhibitor for the Treatment of Iftar-Related Glycemic Excursions in Patients With Type 1 Diabetes on MiniMed™ 780G Advanced Hybrid Closed Loop System
Brief Title: Feasibility of DPP-4 Inhibitor Therapy on Advanced Hybrid Closed Loop System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Prof. of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain Shams University 232212
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Time in Range
MeSH Terms: interventions — Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dipeptidyl peptidase-4 inhibitors (Active Comparator): Dipeptidyl peptidase-4 inhibitors with Iftar meal
  Interventions: Drug: Dipeptidyl peptidase-4 inhibitors
- Control group (No Intervention): No Dipeptidyl peptidase-4 inhibitors intake with Iftar meal

INTERVENTIONS:
Drug: Dipeptidyl peptidase-4 inhibitors — Dipeptidyl peptidase-4 inhibitors with Iftar meal
  Arms: Dipeptidyl peptidase-4 inhibitors

SUMMARY:
Background: Ramadan Iftar meal typically causes glucose excursions. Dipeptidyl peptidase-4 inhibitors increase serum concentrations of glucagon-like peptide-1 and thus, decrease blood glucose levels with low risk of hypoglycemia.

Aim: To investigate the efficacy and safety of vildagliptin as an add-on therapy among adolescents and young adults with type 1 diabetes mellitus (T1DM) on glucose excursions of Iftar Ramadan meals and glycemic metrics during advanced hybrid closed-loop (AHCL) treatment.

DETAILED DESCRIPTION:
Current management of people with type 1 diabetes mellitus (T1DM) on intensive insulin therapy recognizes carbohydrates as the most important determinant of postprandial glycaemia; hence, worldwide guidelines recommend carbohydrates counting for determining pre-prandial insulin doses. Currently, the insulin to carbohydrate ratio (ICR) is frequently used to calculate the meal insulin dose. However, ICRs are considered difficult, ineffective and inaccurate for some patient, with an estimation error of around 20% in adults demonstrating only modest improvements in glycated hemoglobin (HbA1c). This lack of effectiveness and the wide variability using ICRs suggests it should be improved upon.

However, there have been only a few randomized control studies that investigated the efficacy and safety of DPP-4 inhibitors as an add-on drug in patients treated with basal insulin. Therefore, we conducted a one-month randomized control trial to investigate the efficacy and safety of DPP-4 inhibitors as an add-on therapy among adolescents and young adults with T1DM on glucose excursions of Iftar Ramadan meals and glucometrics during AHCL treatment .

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes (T1DM )for at least one year
* patients aged 12-27 years
* patients using MiniMed 780G AHCL system (Medtronic, Northridge, CA, USA) at least 6 months before the study
* patients with minimum daily insulin requirement of more than 8 units
* patients willingness and ability to adhere to the study protocol, access to the internet and a computer system that met requirements for uploading the study pump data.

Exclusion Criteria:

* patients with any microvascular or macrovascular complications
* pregnancy, lactation
* patients who had a point-of-care screening HbA1c >10.0% (86 mmol/mol)
* patients with hypoglycemic unawareness or recurrent severe hypoglycemic episode in the last 6 months prior to recruitment
* patients with recurrent DKA (more than 2 episodes in the previous 6 months).
* patients with any chronic medical condition, current use of medications (other than insulin) that are known to affect blood glucose level.
* patients who had prior adverse reactions to the adjunctive agent

Ages: 12 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
peak postprandial plasma glucose (PPG) level in mg/dl | 4 weeks
  peak postprandial plasma glucose (PPG) level in mg/dl

SECONDARY OUTCOMES:
Time in range % | 4 weeks
  Time in range %

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dyson PA, Twenefour D, Breen C, Duncan A, Elvin E, Goff L, Hill A, Kalsi P, Marsland N, McArdle P, Mellor D, Oliver L, Watson K. Diabetes UK evidence-based nutrition guidelines for the prevention and management of diabetes. Diabet Med. 2018 May;35(5):541-547. doi: 10.1111/dme.13603. PMID 29443421
- [Background] Brazeau AS, Mircescu H, Desjardins K, Leroux C, Strychar I, Ekoe JM, Rabasa-Lhoret R. Carbohydrate counting accuracy and blood glucose variability in adults with type 1 diabetes. Diabetes Res Clin Pract. 2013 Jan;99(1):19-23. doi: 10.1016/j.diabres.2012.10.024. Epub 2012 Nov 10. PMID 23146371
- [Background] Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM, Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL Trial Research Group. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi: 10.1056/NEJMoa1907863. Epub 2019 Oct 16. PMID 31618560
- [Background] Wadwa RP, Reed ZW, Buckingham BA, DeBoer MD, Ekhlaspour L, Forlenza GP, Schoelwer M, Lum J, Kollman C, Beck RW, Breton MD; PEDAP Trial Study Group. Trial of Hybrid Closed-Loop Control in Young Children with Type 1 Diabetes. N Engl J Med. 2023 Mar 16;388(11):991-1001. doi: 10.1056/NEJMoa2210834. PMID 36920756
- [Background] Lakshman R, Boughton C, Hovorka R. The changing landscape of automated insulin delivery in the management of type 1 diabetes. Endocr Connect. 2023 Jul 31;12(8):e230132. doi: 10.1530/EC-23-0132. PMID 37289734
- [Derived] Elbarbary NS, Ismail EAR. Mitigating iftar-related glycemic excursions in adolescents and young adults with type 1 diabetes on MiniMed 780G advanced hybrid closed loop system: a randomized clinical trial for adjunctive oral vildagliptin therapy during Ramadan fasting. Diabetol Metab Syndr. 2023 Dec 7;15(1):257. doi: 10.1186/s13098-023-01232-5. PMID 38057844